CLINICAL TRIAL: NCT01245920
Title: Effects of Bone Graft Placement at Implant Installation on Buccal Plate Stability: A Randomized Controlled Clinical Trial
Brief Title: Effects of Bone Graft Placement at Implant Installation on Buccal Plate Stability
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate number of patients whou could meet inclusion criteria.
Sponsor: Creighton University (Other)
Collaborators: Nebraska Society of Periodontology (Unknown)
Responsible Party: Melissa S. Lang, DDS, MS, Creighton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-15770
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Peri-implant Alveolar Bone Thickness
Keywords: Dental implant; Alveolar bone; Clinical attachment Level

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FDBA + Membrane Group (Experimental): For patients in the FDBA + membrane group, a layer 4 mm thick of cancellous allograft bone (Puros Cancellous, Zimmer Dental inc., Carlsbad, CA) will be placed over the buccal bone in the area of the implant. A resorbable collagen membrane (Bio-Gide, 13 x 25 mm, Osteohealth, Shirley, NY) will be trimmed to extend 5 mm beyond the implant borders and to cover the implant head. Following membrane placement over the bone graft, the gingival flaps will be closed and sutured with 4-0 Vicryl (Ethicon Inc., Sommerville, NJ) with passive tension flap closure.
  Interventions: Biological: DFDBA + Bio-Gide Membrane
- Non-FDBA (Active Comparator): Patients in the non-FDBA group will have gingival flaps closed with the same suturing technique.
  Interventions: Other: Non-FDBA

INTERVENTIONS:
Biological: DFDBA + Bio-Gide Membrane — For patients in the FDBA + membrane group, a layer 4 mm thick of cancellous allograft bone (Puros Cancellous, Zimmer Dental inc., Carlsbad, CA) will be placed over the buccal bone in the area of the implant. A resorbable collagen membrane (Bio-Gide, 13 x 25 mm, Osteohealth, Shirley, NY) will be trimmed to extend 5 mm beyond the implant borders and to cover the implant head. Following membrane placement over the bone graft, the gingival flaps will be closed and sutured with 4-0 Vicryl (Ethicon Inc., Sommerville, NJ) with passive tension flap closure.
  Other Names: Puros bone allograft; Bio-Gide membrane
  Arms: FDBA + Membrane Group
Other: Non-FDBA — Patients in the non-FDBA group will have gingival flaps closed with the same suturing technique.
  Arms: Non-FDBA

SUMMARY:
This randomized clinical trial will involve at least 25 patients who have selected to receive a dental implant to replace a missing tooth. One group will receive the test treatment of a bone graft and a dissolvable membrane at the outer surface of the dental, while the control group will not receive the bone graft and membrane adjacent to the implant.

The following will be measured: bone thickness and height adjacent to implant, inflammation of gum tissue, recession of gum tissue, bleeding, pocket depth, and implant success. Patients will be followed for 1 year, including evaluation time points at 2 weeks, 1 month, 3 and 6 months, and 1 year. Statistical analysis of the data will be conducted.

The hypothesis is that there is no difference with regard to bone thickness, bone height, pocket depth, bleeding, and implant success rate for grafted implant sites compared to non-grafted implant sites.

DETAILED DESCRIPTION:
Our study will include 25 patients. All patients will receive a comprehensive oral evaluation and periodontal examination prior to entry to this study. Patients will be selected on the basis of meeting the inclusion criteria, whose treatment plan is to receive an endosseous dental implant. They will be given oral hygiene instruction at each follow-up appointment. All test and control materials will be strictly controlled by the principal investigator who will maintain all study and patient information in a locked cabinet in a locked room to ensure patient privacy.

Primary Intervention:

Surgical Procedures:

Patients will rinse with 0.12% chlorhexidine gluconate for 60 s before the surgery, and 2 g amoxicillin or 600 mg clindamycin (if allergic to penicillin) will be administered. Sulcular and crestal incisions will be placed in the area of the planned implant. A full-thickness mucoperiosteal flap will be reflected. Surgical placement of an endosseous dental implant (Prima Implant System, Keystone Dental) will be carried out according to manufacturer's recommendation with the use of a surgical template. Following preparation of the osteotomy site to receive the implant, the thickness of the residual buccal bone will be measured and recorded to the nearest 0.5 mm, at approximately 0.5 mm apical to the crest with a caliper. After placement of the implant, the distance between the bony crest and the top of the implant will be measured and recorded to the nearest 1 mm for the buccal aspect of each implant with a periodontal probe (UNC-15). Titanium cover screws will be attached to the implants.

If the patient meets the inclusion criteria (buccal plate thickness is ≥1 mm), the treatment will be selected randomly through a coin toss. Heads indicates the subject will be entered in the FDBA + membrane group. Tails indicates the subject will be entered in the control group (non-FDBA).

Periosteal releasing incisions will be made to adequately mobilize the full-thickness mucoperiosteal flap. For patients in the FDBA + membrane group, a layer 4 mm thick of cancellous allograft bone (Puros Cancellous, Zimmer Dental inc., Carlsbad, CA) will be placed over the buccal bone in the area of the implant. A resorbable collagen membrane (Bio-Gide, 13 x 25 mm, Osteohealth, Shirley, NY) will be trimmed to extend 5 mm beyond the implant borders and to cover the implant head. Following membrane placement over the bone graft, the gingival flaps will be closed and sutured with 4-0 Vicryl (Ethicon Inc., Sommerville, NJ) with passive tension flap closure. Patients in the non-FDBA group will have gingival flaps closed with the same suturing technique. A post-operative periapical radiograph will be exposed of the implant.

Post-operative care will include oral administration of 500 mg amoxicillin 3 times daily for 7 days or 300 mg clindamycin 3 times daily for 7 days. Ibuprofen 600 mg every 8 h for 5 days will be prescribed for analgesics. Patients will be instructed to rinse with 0.12% chlorhexidine gluconate (Peridex, Zila Inc. Pheonix, AZ) twice daily for 1 month. Sutures will be removed 2 weeks post-surgery. Post-surgical evaluations will be provided at 2 weeks, 1 month, 3, and 6 months.

Stage II surgery will be performed 6 months after implant placement using the same flap design as the implant placement surgery. The titanium cover screw will be removed, and replaced with a titanium healing abutment. The distance from the bony crest to the top of the implant will be measured using the same technique described at the implant placement surgery. The buccal bone thickness will be measured by recording the distance from the buccal implant surface to the outer buccal bone crest to the nearest 1 mm using a periodontal probe (UNC-15). Photos of the study site will be taken at each surgical procedure and at each follow-up appointment.

Post-Surgical Clinical Measurements:

The following clinical measurements will be obtained with a plastic periodontal probe at 6 sites at each implant (Colorview, Hu-Friedy, Chicago, IL) and recorded to the nearest millimeter: probing depth, gingival margin position, bleeding on probing, and gingival index. The gingival index will be assessed according to Silness and Loe on a scale of 0-3. Implant mobility will also be assessed using an instrument handle and a finger. The soft tissue clinical measurements will be obtained at the following time periods: 1 month following Stage II surgery and 6 months following Stage II surgery (1 year after implant placement). Final implant abutments and crowns will proceed according to the original treatment plan of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to follow study procedures.
2. Subjects treatment plan includes the placement of at least one endosseous dental implant in the maxillary or mandibular arch.
3. Subjects must present with at least 1 mm buccal bone thickness immediately after surgical placement of endosseous dental implant.
4. Subjects must demonstrate a plaque index of ≤20%.
5. Subjects who can read, understand, and sign an institutional review board approved informed consent.

Exclusion Criteria:

1. Subjects with systemic condition including diabetes mellitus, cancer, human immunodeficiency virus, or bone metabolic disease.
2. Subjects who take corticosteroids, immunosuppressant, bisphosphonates, radiation treatments, and/or chemotherapeutics that could compromise wound healing process.
3. Subjects with acute infectious lesions in the area of study.
4. Subjects under 21 years of age.
5. Subjects with previous failed endosseous dental implant at the site of study.
6. Smokers.
7. Subjects with dehiscence of implant surface > 1 mm immediately after surgical placement of endosseous dental implant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in Buccal Bone Thickness | 6 months
  The buccal bone thickness will be measured by recording the distance from the buccal implant surface to the outer buccal bone crest to the nearest 1 mm using a periodontal probe (UNC-15).

SECONDARY OUTCOMES:
Change in Clinical Attachment Level | 1 year
  The following clinical measurements will be obtained with a plastic periodontal probe at 6 sites at each implant (Colorview, Hu-Friedy, Chicago, IL) and recorded to the nearest millimeter: probing depth and gingival margin position

CONTACTS AND LOCATIONS:
Overall Officials: Melissa S Lang, DDS, MS, Principal Investigator — Creighton University School of Dentistry
Locations (1):
- Creighton University School of Dentistry, Omaha, Nebraska, United States